CLINICAL TRIAL: NCT03577626
Title: Randomized, Open-labeled, Single Dosing Study to Assess Food Effect on the Pharmacokinetics of Hemay005 in Healthy Volunteers
Brief Title: A Food Effect Study to Assess Pharmacokinetics of Hemay005 in Healthy Volunteers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Hemay Bio-Tech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM005PS1S02
Record Dates: First submitted 2018-06-22; First posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-06

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Hemay005

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemay005 Fast (Experimental)
  Interventions: Drug: Hemay005
- Hemay005 Fed (Experimental)
  Interventions: Drug: Hemay005

INTERVENTIONS:
Drug: Hemay005 — Hemay005 tablets will be taken orally in dose of 52.5mg at fasted dosing on period one followed by fed dosing on period two.
  Arms: Hemay005 Fast
Drug: Hemay005 — Hemay005 tablets will be taken orally in dose of 52.5mg at fed dosing on period one followed by fasted dosing on period two
  Arms: Hemay005 Fed

SUMMARY:
The purpose of this study is to evaluate the effect of food on the PK of a single dose of 52.5 mg Hemay005 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. healthy subjects aged 18 to 60 years, male and female volunteers;
2. male Bodyweight（BW）≥ 50kg, female Bodyweight（BW）≥ 45kg, Body mass index (BMI) in 18-28 (including upper and lower limit of the range);
3. All male subjects must agree and commit to the use of a reliable contraceptive regimen(including vasoligation, abstinence, using a condom) for the duration of the study(from screening until 6 months after the last dose), Female participants with a negative pregnancy test (serum) at both the screening visit and at Day-1, Female subjects and female partners of male subjects must agree and commit to the use of a reliable contraceptive regimen ( oral contraceptive medications or non-oral contraceptive medications) for the duration of the study(from screening until 6 months after the last dose);
4. Ability to understand and be willing to sign a written informed consent before study entry;
5. Subjects would have good communication with the investigator and could comply with protocol.

Exclusion Criteria:

1. A history of clinically severe gastrointestinal, hepatic, renal, cardiovascular, dermatological, immunological, respiratory, endocrine, oncological, neurological, metabolic, psychiatric disease or haematological disorders;
2. Have a known history of hypersensitivity to any medicine or food, or allergy to the test article or any of the excipient of the test article;
3. Have a gastrointestinal, hepatic or renal condition that may influence drug absorption or metabolism;
4. A history of chronic infection (ie, tuberculosis);
5. A medical history of any clinically significant medical disease or surgery within 4 weeks of the screening;
6. Clinically significant laboratory abnormal results at screening or prior to the first dose of study drug;
7. Clinically significant abnormal 12-lead ECG or vital signs ( systolic pressure <90 mmHg or >140 mmHg, diastolic pressure <50 mmHg or >90 mmHg; radial pulse rate <50 bpm or >100 bpm);
8. Positive blood screen for human immunodeficiency virus (HIV antibody), hepatitis B virus surface antigen, or hepatitis C virus antibody at screening;
9. Recent history of frequent alcohol consumption, defined by average intake of greater than 14 units of alcohol per week (1 unit = 360 mL beer or 45 mL of spirits with 40% alcohol content, or 150 mL wine), Participants who are unable to abstain from smoking during the study or quitting smoking for less than 3 months;
10. Positive urine screen for drug and cigarettes, positive breath test for alcohol;
11. Subjects who use soft drugs (ie marijuana )within 3 months of the screening and entire study duration or hard drugs (ie cocaine, phencyclidine ) within 1 year of the screening and entire study duration;
12. Dietary habits or food intolerances which will interfere with the requirements for participants to consume a standardised diet whilst confined to the clinical unit;
13. Participants who eat special food (Including grapefruit and/or Xanthine diet) for 14 days prior to dosing or any caffeine containing food or drinks, i.e. chocolate for 48 hours prior to dosing or drinking alcohol for 24 hours prior to dosing and not will stop to intake above food and drinks;
14. Use of any drug that inhibits or induces hepatic metabolism of drugs within 30 days of planned study drug administration and entire study duration (e.g. inducers: barbiturates, carbamazepine, rifampicin, phenytoin, glucocorticoid and omeprazole; inhibitors - SSRI antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedatives and hypnotics, verapamil, fluoroquinolones and antihistamines);
15. Participant who received any medicine within 14 days of the initial dose of study drug;
16. Have received other clinical trials treatment within 3 months prior to study;
17. Participants who have donated of blood (>400 mL) within 4 weeks of the study, or plan to donate of blood during of the study and 4 weeks after the study;
18. Subjects cannot complete the study due to other reasons or by the investigator's judgment;
19. Pregnancy or lactating females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-10-10 (Estimated); Primary Completion 2018-11-10 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Cmax | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 ,72hours post-dose on day 1 and day 8
  Maximum observed plasma concentration
Tmax | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 ,72hours post-dose on day 1 and day 8
  Time of maximum concentration
AUCt | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 ,72hours post-dose on day 1 and day 8
  Area under the plasma concentration-time curve from time zero to the last quantifiable concentration
AUC∞ | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 ,72hours post-dose on day 1 and day 8
  Area under the plasma concentration-time curve from time zero extrapolated to infinity
t1/2 | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 ,72hours post-dose on day 1 and day 8
  Terminal elimination half-life
CL/F | pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 24, 36, 48 ,72hours post-dose on day 1 and day 8
  Apparent total plasma clearance

SECONDARY OUTCOMES:
Number of participants with adverse events, serious adverse events | Day 1 up to Day 11±3

CONTACTS AND LOCATIONS:
Overall Officials: Hongyun Wang, Doctor, Principal Investigator — Peking Union Medical College Hospital